CLINICAL TRIAL: NCT02071238
Title: Factors Affecting Risk Recall in Open Carpal Tunnel Release Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Bezuhly (Other)
Responsible Party: Sponsor-Investigator, Michael Bezuhly, Plastic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CDHA-RS/2014-244
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Carpal Tunnel
Keywords: Carpal tunnel; Carpal tunnel release; Risk Recall; Patient satisfaction; Pamphlet; Brochure
MeSH Terms: conditions — Median Neuropathy; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pamphlet (Experimental): Patient group that will receive a written pamphlet outlining the risks of surgery as discussed in consultation.
  Interventions: Behavioral: Pamphlet
- No pamphlet, individual (No Intervention): Patient group that will not receive a written pamphlet outlining the risks of surgery as discussed in consultation.
- Group Consultation (Experimental): Patient group that will receive informed consent discussion in a group-format.
  Interventions: Behavioral: Group Consultation

INTERVENTIONS:
Behavioral: Pamphlet — Written pamphlet outlining the risks of surgery as discussed in consultation.
  Arms: Pamphlet
Behavioral: Group Consultation — Informed consent discussion in group-format
  Arms: Group Consultation

SUMMARY:
Understanding of an operation and its risks has been shown to give patients more realistic expectations, increase cooperation and result in higher satisfaction. Traditionally, informed consent for surgical procedures involve a discussion between the surgeon and the patient, but many patients easily forget the details of these talks. The investigators wish to investigate if providing a written pamphlet along with the standard oral discussion improves patients' ability to remember the details of the operation, improving the quality of the informed consent process.

In addition, we will test whether a group consultation format provides a model for large-volume, low-variation, low-urgency surgery without reducing ability to recall risks of surgery or overall satisfaction.

DETAILED DESCRIPTION:
Objective of this study The investigators' study objectives are to see if additionally providing a written document along with the discussion of surgical risks improves risk recall for patient seen in consultation for open carpal tunnel release, and if this has any effect on overall satisfaction after the procedure.

To accomplish this goal, the investigators intend to provide patients with a written document outlining the same risks as are discussed in consultation and investigate if their recall of the risks is improved compared to patients who receive discussion alone. The investigators will also see whether risk recall is affected if patients participate in a group format informed consent discussion compared to a standard individual discussion. The investigators propose to do this as a two-part prospective randomized control trial of patients who are new referrals to the Halifax Infirmary Plastic Surgery Clinic.

Background The informed consent process The risks and benefits of an operation or procedure are typically discussed as part of the informed consent process for an initial surgical consultation. Informed consent is a legal requirement for surgery and is based on the components of disclosure, comprehension, competence and voluntary choice. Despite this, patients are often unable to recall the specific risks that were reviewed. Additionally, failure to understand the possible risks and failure of communication are more common reasons for patients to seek legal action. Patients have historically reported that they wished they had received more information about their operation prior to surgery.

Increased understanding of a procedure and its risks has been shown to give patients more realistic expectations, increase cooperation and result in higher satisfaction. Traditionally, obtaining informed consent for surgical procedures has involved an oral discussion, but this may be insufficient as oral information tends to be poorly retained.

Previous research in the field of otolaryngology has shown that written documentation in addition to oral discussion increases recall of both general knowledge of a procedure and of the specific risks of a procedure. Siau et al. (2010) found that this effect was even more pronounced for recall of the risks associated with the operation and that subjectively patients were found to be happy to have received a pamphlet and found it helpful. Early research into this subject in general surgery suggested that the optimal time to provide additional information regarding a procedure is at the time of the initial consultation or at least one week prior to surgery.

The investigators' research is important as it could show that providing a written document in conjunction with the standard oral discussion improves patients' risk recall in the informed consent process for open carpal tunnel surgery. In addition, the investigators wish to look into whether this in turn increases satisfaction with the procedure. Though past research has drawn a link between comprehension and satisfaction, very little research has been conducted specifically on this topic. In the future this research could be extended to other surgical practices.

Due to large volumes of patients requiring open carpal tunnel release, wait times following referral can vary from 30 to 151 days in Nova Scotia, with an average wait time of 59 days (Patient Access Registry NS, July-September 2013). While open carpal tunnel release surgery is a very brief procedure with an extremely low rate of post-operative complications (Ono et al., 2010), the presurgical consultation with each patient takes a large proportion of the time spent by both patient and surgeon addressing the disease. To address a similar problem involving extensive information required prior to surgery, the UHN breast reconstruction program in Toronto is in the process of piloting an educational group intervention, which includes seminar-style lectures and group discussion, in order to improve shared decision making in women undergoing post-mastectomy breast reconstruction (Platt et al., 2013). We seek to implement a similar program for patients scheduled to undergo open carpal tunnel release.

According to the Weiss model of medical stigma (Weiss et al., 2006), Carpal Tunnel Syndrome could be considered a disease with minimal stigma attached. As one would correspondingly expect, when offered the opportunity to participate in a group seminar style presurgical consult, many patients have expressed a positive opinion and willingness to participate.

If there are no differences between risk recall or general satisfaction in patients who are part of a group consultation compared to a traditional consult, group consultation may be a viable tool to shorten wait times for patients undergoing specific kinds of medical and surgical procedures.

Hypothesis The investigators are testing whether providing a written document in conjunction with the standard oral discussion improve patients' risk recall in the informed consent process for open carpal tunnel release and increase patients' subjective satisfaction with their operation. In addition, the investigators will test whether a group consultation format provides a model for large-volume, low-variation, low-urgency surgery without reducing ability to recall risks of surgery or overall satisfaction.

Patient Selection

The investigators study will be a two-part prospective randomized study, each of 100 consecutive patients being seen for open carpal tunnel release consultation at the Halifax Infirmary. Inclusion criteria will be:

The sample size was chosen based on previous studies investigating risk recall and a power calculation with the hypothesis of a mean of 4 items recalled, a standard deviation of 2.5 (alpha 0.05, beta 0.95), giving us a sample size given our hypothesis (n = 40 per study group).

ELIGIBILITY:
Inclusion Criteria:

* Referral to the Halifax Infirmary plastic surgery clinic for consultation for open carpal tunnel release

Exclusion Criteria:

* Age less than 16 years
* Inability to fluently communicate in English
* Discussion of additional procedures
* Prior open (not percutaneous) hand surgery
* Inability to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of risks recalled | 2-3 weeks
  Number of risks discussed at time of initial visit that are remembered by the patient at a 2 week follow up phone call.

SECONDARY OUTCOMES:
Patient Satisfaction | 3 months
  Patients' perceived satisfaction, as measured by a visual-analogue scale rating their satisfaction with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bezuhly, MD MSc SM, Principal Investigator — 902-470-8168
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Lavelle-Jones C, Byrne DJ, Rice P, Cuschieri A. Factors affecting quality of informed consent. BMJ. 1993 Apr 3;306(6882):885-90. doi: 10.1136/bmj.306.6882.885. PMID 8490411
- [Background] Nadeau DP, Rich JN, Brietzke SE. Informed consent in pediatric surgery: Do parents understand the risks? Arch Otolaryngol Head Neck Surg. 2010 Mar;136(3):265-9. doi: 10.1001/archoto.2010.5. PMID 20231645
- [Background] Schenker Y, Fernandez A, Sudore R, Schillinger D. Interventions to improve patient comprehension in informed consent for medical and surgical procedures: a systematic review. Med Decis Making. 2011 Jan-Feb;31(1):151-73. doi: 10.1177/0272989X10364247. Epub 2010 Mar 31. PMID 20357225
- [Background] Leclercq WK, Keulers BJ, Scheltinga MR, Spauwen PH, van der Wilt GJ. A review of surgical informed consent: past, present, and future. A quest to help patients make better decisions. World J Surg. 2010 Jul;34(7):1406-15. doi: 10.1007/s00268-010-0542-0. PMID 20372902
- [Background] Kessler TM, Nachbur BH, Kessler W. Patients' perception of preoperative information by interactive computer program-exemplified by cholecystectomy. Patient Educ Couns. 2005 Nov;59(2):135-40. doi: 10.1016/j.pec.2004.10.009. PMID 16257617
- [Background] Siau D, List RJ, Hussin N, Woolford TJ. Do printed information leaflets improve recall of the procedure and risks in adult tonsillectomy? How we do it. Clin Otolaryngol. 2010 Dec;35(6):503-6. doi: 10.1111/j.1749-4486.2010.02227.x. No abstract available. PMID 21199416
- [Background] Hong P, Makdessian AS, Ellis DA, Taylor SM. Informed consent in rhinoplasty: prospective randomized study of risk recall in patients who are given written disclosure of risks versus traditional oral discussion groups. J Otolaryngol Head Neck Surg. 2009 Jun;38(3):369-74. PMID 19476770
- [Background] Ono S, Clapham PJ, Chung KC. Optimal management of carpal tunnel syndrome. Int J Gen Med. 2010 Aug 30;3:255-61. doi: 10.2147/ijgm.s7682. PMID 20830201
- [Background] Platt J, Baxter N, Jones J, Metcalfe K, Causarano N, Hofer SO, O'Neill A, Cheng T, Starenkyj E, Zhong T. Pre-consultation educational group intervention to improve shared decision-making in postmastectomy breast reconstruction: study protocol for a pilot randomized controlled trial. Trials. 2013 Jul 6;14:199. doi: 10.1186/1745-6215-14-199. PMID 23829442
- [Background] Weiss MG, Ramakrishna J, Somma D. Health-related stigma: rethinking concepts and interventions. Psychol Health Med. 2006 Aug;11(3):277-87. doi: 10.1080/13548500600595053. PMID 17130065